CLINICAL TRIAL: NCT07240545
Title: The Effectiveness of Chewing Gum for Reducing Cigarette Consumption and Promoting Smoking Cessation: A Pilot Randomized Controlled Trial
Brief Title: Xylitol Gum for Promoting Smoking Cessation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof. Wang Man-Ping, Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Chew 2 quit
Record Dates: First submitted 2025-11-16; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Smoking Cessation; Health Promotion
Keywords: Xylitol gum; Smoking cessation; Hybrid type 1 effectiveness-implementation design
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants assigned to the intervention group will receive a 3-month behavioral intervention comprising a 4-week xylitol gum aligned with 12 weeks of instant reminder message support.
  Interventions: Behavioral: Brief smoking cessation advice; Behavioral: Warning leaflet; Behavioral: Self-help smoking cessation booklet; Behavioral: 4-week xylitol gum intervention; Behavioral: Instructional leaflet; Behavioral: 12-week instant message support
- Control group (Active Comparator): Participants in the control group will receive brief SC advice and a SC information booklet at baseline, which had been routinely used in our previous trials.
  Interventions: Behavioral: Brief smoking cessation advice; Behavioral: Warning leaflet; Behavioral: Self-help smoking cessation booklet

INTERVENTIONS:
Behavioral: Brief smoking cessation advice — Brief smoking cessation advice guided by the validated AWARD model (Assess, Warning, Advice, Refer, and Do-it-again).
Behavioral: Warning leaflet — The warning leaflet contains pictorial depictions of the adverse health effects of smoking.
Behavioral: Self-help smoking cessation booklet — The self-help smoking cessation booklet includes commonly used smoking cessation strategies.
Behavioral: 4-week xylitol gum intervention — Participants in the intervention group will receive 4 packs of xylitol gum (approximately US $2 per pack) at baseline and will be encouraged to use it when they experience cravings.
  Arms: Intervention group
Behavioral: Instructional leaflet — The instructional leaflet includes the potential benefits of xylitol gum for smoking cessation, recommended timing and dosage for use, and appropriate disposal of used gum.
  Arms: Intervention group
Behavioral: 12-week instant message support — Approximately 24 reminder messages (two per week), developed based on the Love and Care Approach framework, will be delivered over the 12-week period to reinforce motivation and adherence.
  Arms: Intervention group

SUMMARY:
The goal of this clinical trial is to learn if 4-week xylitol gum intervention works to promote smoking cessation in daily smokers. It will also learn about the feasibility and acceptability of using xylitol gum. The main questions it aims to answer are:

（1）Does xylitol gum help to reduce cigarette consumption and promote smoking cessation?

Researchers will compare 4-week xylitol gum intervention to the brief advice to see if xylitol gum works to promote smoking cessation.

Participants in the intervention group will receive a 3-month behavioral intervention comprising a 4-week xylitol gum aligned with 12 weeks of instant reminder message support.

DETAILED DESCRIPTION:
This study aims to evaluate the feasibility, acceptability, and preliminary effectiveness of a proactive smoking cessation intervention using xylitol chewing gum. Eligible participants will be Hong Kong residents aged ≥18 years who (1) have smoked at least one cigarette per day in the past 3 months; (2) can communicate in Cantonese (including reading Chinese); (3) express an intention to quit or reduce smoking; (4) are able to use instant messaging tools (e.g., WhatsApp); and (5) regularly chew gum or are willing to use chewing gum for smoking reduction.

A total of 134 participants will be recruited from community settings, including public housing estates across Hong Kong's 18 districts, community and university smoking hotspots, referrals from other smoking cessation programmes, and social media promotions (Facebook and Instagram). The study will adopt a hybrid type I effectiveness-implementation design. Participants will be followed up at 1, 3, and 6 months post-enrolment via telephone, following CONSORT guidelines, to assess cigarette reduction and cessation outcomes.

All participants will receive brief smoking cessation advice at baseline using the AWARD model (Ask/Assess, Warn, Advise, Refer, and Do-it-again), accompanied by a health warning leaflet and a smoking cessation information booklet.

Interventions are as follows:

Chewing gum group (intervention): Participants will receive 4 packs of xylitol gum at baseline and up to 24 packs throughout the 12-week intervention. Approximately 24 reminder messages (two per week), developed based on the Love and Care Approach framework, will be delivered via instant messaging to reinforce motivation and adherence.

Unassisted quitting group (control): Participants will receive brief advice only at baseline.

To explore user experience and acceptability, semi-structured qualitative interviews will be conducted with 20 intervention-group participants to understand their perceptions and experiences with xylitol gum use.

The primary outcome is biochemically validated smoking abstinence at 6 months, defined as exhaled carbon monoxide <4 ppm and salivary cotinine <30 ng/mL.

ELIGIBILITY:
Inclusion Criteria:

* Residents of Hong Kong aged 18 or above who smoke at least 1 cigarette per day over the past 3 months
* Have the habit of chewing gum or are willing to use chewing gum
* Can communicate in Cantonese (including reading Chinese)
* Express an intention to quit or reduce smoking
* Capable of using instant messaging tools (e.g., WhatsApp, WeChat) for communication

Exclusion Criteria:

* Have communication barriers (either physical or cognitive)
* Currently participating in other smoking cessation programs or services

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2025-11-24 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Biochemically validated smoking abstinence | 6-month follow-up
  Verified by exhaled carbon monoxide <4 ppm and salivary cotinine <30 ng/ml

SECONDARY OUTCOMES:
Biochemically validated smoking abstinence | 3-month follow-up
  Verified by exhaled carbon monoxide <4 ppm and salivary cotinine <30 ng/ml
Self-report 7-day point-prevalence abstinence | 1-, 3-, and 6-months follow-ups
  By asking a question, "Have you smoked (even a puff) during the past 7 days?"
Smoking reduction | 1-, 3-, and 6-months follow-ups
  Defined by a reduction of≥50% in daily cigarette consumption compared with baseline.
Quit attempt | 1-, 3-, and 6-months follow-ups
  By asking a question, "Have you attempted to stop smoking completely for at least 24 hours in the past 7 days?"

OTHER OUTCOMES:
Number of pieces of xylitol gum used | 1- and 3-month follow-ups
  Total daily count used during the intervention period
Frequency of using xylitol gum | 1- and 3-month follow-ups
  Average number of chewing episodes per day.
Duration of use | 1- and 3-month follow-ups
  Average time spent chewing each piece.

CONTACTS AND LOCATIONS:
Overall Officials: Man Ping Wang, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- School of Nursing, The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No